CLINICAL TRIAL: NCT05476991
Title: Reducing Inflammation in Ischemic Stroke With Colchicine, and Ticagrelor in High-risk Patients-extended Treatment in Ischemic Stroke
Brief Title: Evaluation of Low Dose Colchicine and Ticagrelor in Prevention of Ischemic Stroke in Patients With Stroke Due to Atherosclerosis
Acronym: RIISC-THETIS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: APHP211055
Record Dates: First submitted 2022-07-25; First posted 2022-07-27 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-06

CONDITIONS: Stroke; Stroke, Ischemic; Atherosclerosis; Myocardial Infarction; Coronary Syndrome; TIA; Cardiac Disease; Cerebral Infarction
Keywords: Stroke; Colchicine; Atherosclerosis; Aspirin; Ticagrelor
MeSH Terms: conditions — Stroke; Ischemic Stroke; Atherosclerosis; Myocardial Infarction; Angina, Unstable; Heart Diseases; Cerebral Infarction | interventions — Colchicine; Ticagrelor; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Colchicine + Ticagrelor (Experimental)
  Interventions: Drug: Colchicine 0.5 MG; Drug: Ticagrelor 90mg
- Colchine + Aspirine (Experimental)
  Interventions: Drug: Colchicine 0.5 MG; Drug: Aspirin 75-300mg
- SOC + Ticagrelor (Experimental)
  Interventions: Drug: Ticagrelor 90mg
- SOC + Aspirine (Active Comparator)
  Interventions: Drug: Aspirin 75-300mg

INTERVENTIONS:
Drug: Colchicine 0.5 MG — Colchicine is a medication used to treat gout and Behçet's disease. In gout, it is less preferred to NSAIDs or steroids. Other uses for colchicine include the management of pericarditis and familial Mediterranean fever.
  Arms: Colchicine + Ticagrelor; Colchine + Aspirine
Drug: Ticagrelor 90mg — Ticagrelor, sold under the brand name Brilinta among others, is a medication used for the prevention of stroke, heart attack and other events in people with acute coronary syndrome, meaning problems with blood supply in the coronary arteries. It acts as a platelet aggregation inhibitor by antagonising the P2Y 12 receptor.
  Other Names: Brilinta
  Arms: Colchicine + Ticagrelor; SOC + Ticagrelor
Drug: Aspirin 75-300mg — Also known as Aspirin, acetylsalicylic acid (ASA) is a commonly used drug for the treatment of pain and fever due to various causes. Acetylsalicylic acid has both anti-inflammatory and antipyretic effects. This drug also inhibits platelet aggregation and is used in the prevention of blood clots stroke, and myocardial infarction (MI).
  Other Names: Acetylsalicylic acid
  Arms: Colchine + Aspirine; SOC + Aspirine

SUMMARY:
REDUCING INFLAMMATION IN ISCHEMIC STROKE WITH COLCHICINE, AND TICAGRELOR IN HIGH-RISK PATIENTS-EXTENDED TREATMENT IN ISCHEMIC STROKE.

DETAILED DESCRIPTION:
Our main hypothesis is that low-dose colchicine (0.5 mg/day) on top of best medical care, in patients with an ischemic stroke with ipsilateral atherosclerotic stenosis, will reduce the risk of major vascular events after 36-60 months of treatment as compared to no colchicine.

Our second main hypothesis, tested in 2x2 factorial design, is that ticagrelor 90 mg bid in the same patients, will reduce the long-term risk of major vascular events (after 36-60 months of treatment) as compared to aspirin 75-300 mg/day.

ELIGIBILITY:
Inclusion criteria:

Patient should have the following:

Patient with:

1. Cerebral infarction (CI) proven by neuro-imaging (MRI or head-CT), immediately once the neurologic deficit is stabilized (investigator judgement) if the patient was on antiplatelet agent monotherapy after the qualifying event, or after 21 days if the patient was on clopidogrel plus aspirin after the qualifying event, or after 21 to 30 days if the patient was on ticagrelor plus aspirin after the qualifying event (TIA with documented ischemic lesion (MRI or CT) in the appropriate area corresponding to the symptoms will be considered CI, following the current definition)
2. Or TIA lasting more 10 minutes or more (with motor symptoms or aphasia/dysarthria or visual defect), with total resolution and no brain lesion on neuro-imaging (TIA) and with ipsilateral carotid stenosis that was revascularized (endarterectomy or stenting) or with ipsilateral, potentially causal intracranial stenosis ≥70%) if the patient was on antiplatelet agent monotherapy after the qualifying event, or after 21 days if the patient was on clopidogrel plus aspirin after the qualifying event, or after 21 to 30 days if the patient was on ticagrelor plus aspirin after the qualifying event
3. and documented atherosclerotic stenosis:

   1. presence of carotid atherosclerotic stenosis (on the basis of carotid duplex, CTA, MRA, XRA - only the report will be required to document atherosclerotic disease) ipsilateral to the cerebral ischemic symptoms (stenosis defined by luminal narrowing ≥30%, judgement of the investigator)
   2. or presence of atherosclerotic stenosis of another cerebral artery (documented vertebral artery stenosis, basilar artery stenosis, other intracranial artery stenosis) ipsilateral to the ischemic area (stenosis defined by luminal narrowing ≥30%, judgement of the investigator)
   3. or presence of atherosclerotic disease of the aortic arch with a plaque ≥4mm in thickness with or without superimposed thrombus, or a plaque <4 mm with a superimposed mobile thrombus (detected by transesophageal echocardiography or CT angiography)
4. with no clear indication of colchicine treatment (gout, Mediterranean fever) and with an indication to long-term antiplatelet therapy (no clear indication to oral anticoagulant)
5. age equal or above 18
6. Rankin score less than ≤4 (ranges from 0 to 6, with 0 indicating no symptoms, 1 no disability, 2 to 3 needing some help with daily activities, 4 to 5 dependent or bedridden, and 6 death),
7. fully informed and signed inform consent
8. with social security number.
9. medical examination before the participation to the research
10. Under contraception in case of childbearing potential (highly effective: 1) combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation et 2) progestogen-only).
11. Pregnancy test for women of childbearing potential

Exclusion Criteria:

1. Colchicine treatment needed (e.g., gout, Mediterranean fever)
2. Hypersensitivity to ticagrelor or any of the excipients.
3. Hypersensitivity to colchicine or any of the excipients.
4. Major digestive disorders (chronic diarrhea, inflammatory disease of the digestive tract as uncontrolled ulcerative colitis or active Crohn disease)
5. Immunosuppression, medullary aplasia
6. Active chronic inflammatory disease, chronic active infection, evolving cancer
7. Hemodynamic instability (need for amines for more than 24 hours, circulatory assistance)
8. A recent severe sepsis (7 days) or all recent acute reaches
9. Chronic treatment (for more than 6 months) with corticosteroids or NSAIDs (or repeated high-dose intake for less than 7 days).
10. Anticipated concomitant oral or intravenous therapy with strong CYP3A4 inhibitors or CYP3A4 substrates than cannot be stopped for the course of the course of this study
11. CI/TIA due to arterial dissection (as documented following the judgment of the investigator) or due to cardiac source of embolism without documented atherosclerotic disease (e.g., mitral stenosis or endomyocardial fibrosis, endocarditis) a patient with atrial fibrillation, or with a history of myocardial infarction, or with calcified aortic stenosis will be eligible if the above inclusion criteria are also met]
12. Indication to long-term oral anticoagulant treatment (e.g., atrial fibrillation)
13. Symptomatic hemorrhagic stroke (the mere presence of asymptomatic cerebral hemosiderin deposits -so called "microbleedings" - on gradient echo imaging is not an exclusion criteria)
14. Active pathological bleeding
15. Uncontrolled hypertension (investigator judgement)
16. Follow-up visit impossible or anticipated bad compliance.
17. Intercurrent disease that may interfere with evaluation of the primary end-point or that may prevent follow-up study visits..
18. Anticipated pregnancy at time of enrollment in the study
19. Breastfeeding woman
20. Patients participating in another pharmaco therapeutic program with an experimental therapy that is known to affect the ticagrerlor, colchicine or aspirine therapy.
21. Leukopenia <3000/μl
22. Patients with severe renal impairment (creatinine clearance < 30 ml/min)
23. Patients with severe hepatic impairment
24. Prohibited treatments: All treatments contraindicated during the use of colchicine and/or ticagrelor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2800 (Estimated)
Dates: Start 2023-05-17 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with nonfatal ischemic stroke | 36 months
  Sudden onset of focal neurologic symptoms related to impaired cerebral circulation. ASCOD phenotyping will be used. TIAs will not be part of strokes. However, any focal neurologic symptoms associated with positive DWI or hypodensity on the CT scan in an appropriate area in relation with these symptoms will be considered a cerebral infarction and be part of "strokes".
Number of Participants with undetermined stroke | 36 months
  Sudden onset of focal neurologic symptoms related to impaired cerebral circulation. ASCOD phenotyping will be used. TIAs will not be part of strokes. However, any focal neurologic symptoms associated with positive DWI or hypodensity on the CT scan in an appropriate area in relation with these symptoms will be considered a cerebral infarction and be part of "strokes".
Number of Participants with nonfatal myocardial infarction | 36 months
  * Fatal or nonfatal myocardial infarction (OMS.AHA/ACC definition)
    o Clinical symptoms + elevated troponin
  * Silent myocardial infarction following universal definition
Number of Participants with urgent coronary or carotid revascularization following new symptoms | 36 months
  Revascularization Procedure
  * Coronary : Angioplasty or stenting or CABG
  * Carotid : angioplasty or stenting, surgical endarterectomy
  * Peripheral: angioplasty or stenting including aorta, surgical by-pass or endarterectomy of a peripheral artery.
Number of Participants with vascular death including sudden death | 36 months
  - Vascular death
  * Death due to cardiac or vascular cause
  * Death due to systemic hemorrhage
  * Death due to pulmonary embolism
  * Sudden death: death occurring within 24 hours, unexpected in a patient in apparent healthy condition or condition that was stable or improved
  * Death without documented nonvascular cause
  * Fatal stroke: death occurring within 30 days of stroke onset (whether ischemic or hemorrhagic).

SECONDARY OUTCOMES:
Number of Participants with recurrent fatal and nonfatal ischemic stroke | 36 months
Number of Participants with urgent carotid revascularization following a new transient ischemic attack with negative neuro-imaging | 36 months
Number of Participants with fatal and nonfatal myocardial infarction | 36 months
Number of Participants with fatal and nonfatal myocardial infarction or urgent coronary revascularization following a new acute coronary syndrome | 36 months
Number of Participants with vascular death | 36 months
Number of Participants with any stroke or TIA | 36 months
  A TIA is defined by sudden onset of neurologic symptoms presumed of ischemic origin, with total resolution, being clearly related to focal cerebral or retinal involvement, and with negative neuro-imaging in the cerebral area corresponding to the symptoms. TIA diagnosis must be confirmed by a neurologist, based on clinical and negative neuro-imaging evaluation (MRI with DWI is recommended).
Number of Participants with major coronary events | 36 months
Number of Participants with any coronary end-points (MI, hospitalization for recurrent ACS, coronary revascularization procedure urgent or elective, fatal coronary event) | 36 months
  ACS: Acute Coronary Syndrome
Number of death participant (any death) | 36 months
Number of Participant with all revascularization procedures (coronary, carotid, peripheral) | 36 months
Number of Participants with Carotid revascularization | 36 months

CONTACTS AND LOCATIONS:
Locations (1):
- URC Lariboisière-Fernand Widal-Saint Louis, Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No